CLINICAL TRIAL: NCT01878214
Title: Effective Communication Strategies for Promoting Smoking Cessation in Carpenters
Brief Title: Promoting Smoking Cessation in Carpenters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201110075; R21CA161169 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-06-14 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Smoking Cessation; Health Behavior; Cancer
Keywords: Health communication; Smoking cessation; Health behavior; Construction industry; Audience segmentation
MeSH Terms: conditions — Smoking Cessation; Health Behavior; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Targeted messaging
  Interventions: Behavioral: Targeted messaging; Behavioral: Standard messaging
- Control group (Active Comparator): Standard messaging
  Interventions: Behavioral: Standard messaging

INTERVENTIONS:
Behavioral: Targeted messaging — 6 targeted mailed messages and 6 booster text messages
  Arms: Intervention group
Behavioral: Standard messaging — 1 informational letter

SUMMARY:
The purpose of this study is to test an innovative and sustainable intervention to increase participation in a union-sponsored smoking cessation program among carpenters and floor layers. The investigators will conduct a randomized controlled trial comparing targeted messaging versus standard messaging. All subjects will receive information about the free, union-sponsored smoking cessation program. Subjects randomized to the intervention group will receive additional targeted materials to encourage enrollment in the union's smoking cessation program. The intervention will include monthly mailed and text messages. The investigators hypothesize that subjects who receive targeted messages will be more likely to enroll in the union-sponsored smoking cessation program, be more likely to show change in readiness to quit smoking, and be more likely to quit smoking compared to subjects who receive only standard messaging.

DETAILED DESCRIPTION:
Specific Aim 1: Develop targeted health messages based on audience segmentation to encourage smokers to enroll in a comprehensive union-sponsored smoking cessation program.

We will craft six specific health messages that appeal to four different audience segments: workers under 30 years old without children, workers under 30 with children, workers 30 years old or older without children, and workers 30 or older with children.

Specific Aim 2: Conduct a randomized controlled trial of targeted messaging based on audience segmentation versus standard smoking cessation messaging.

After conducting baseline surveys with union carpenters and floor layers, we will randomize current smokers (smoked within the last 30 days) into either the intervention or control group.

* Control subjects will receive one standard mailing informing them about the free smoking cessation program available to union members.
* Intervention subjects will receive the standard mailing in addition to six targeted smoking cessation messages delivered monthly by mail to their homes. Messages will be specific to one of four audience segments determined by age and parental status. In addition to a segment-specific anti-smoking message, each mailing will have contact information for the union smoking cessation program. Intervention subjects who consented to text messaging will also receive one booster text message each month with a shortened targeted message.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (smoked cigarettes within the last 30 days)
* Eligible for union health benefits

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Evanoff, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Barbeau EM, Krieger N, Soobader MJ. Working class matters: socioeconomic disadvantage, race/ethnicity, gender, and smoking in NHIS 2000. Am J Public Health. 2004 Feb;94(2):269-78. doi: 10.2105/ajph.94.2.269. PMID 14759942
- [Background] Barbeau EM, Li Y, Calderon P, Hartman C, Quinn M, Markkanen P, Roelofs C, Frazier L, Levenstein C. Results of a union-based smoking cessation intervention for apprentice iron workers (United States). Cancer Causes Control. 2006 Feb;17(1):53-61. doi: 10.1007/s10552-005-0271-0. PMID 16411053
- [Background] Bock B, Graham A, Sciamanna C, Krishnamoorthy J, Whiteley J, Carmona-Barros R, Niaura R, Abrams D. Smoking cessation treatment on the Internet: content, quality, and usability. Nicotine Tob Res. 2004 Apr;6(2):207-19. doi: 10.1080/14622200410001676332. PMID 15203794
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Fagerstrom KO, Schneider NG. Measuring nicotine dependence: a review of the Fagerstrom Tolerance Questionnaire. J Behav Med. 1989 Apr;12(2):159-82. doi: 10.1007/BF00846549. PMID 2668531
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Ham DC, Przybeck T, Strickland JR, Luke DA, Bierut LJ, Evanoff BA. Occupation and workplace policies predict smoking behaviors: analysis of national data from the current population survey. J Occup Environ Med. 2011 Nov;53(11):1337-45. doi: 10.1097/JOM.0b013e3182337778. PMID 21988795
- [Background] Kreuter MW, Wray RJ. Tailored and targeted health communication: strategies for enhancing information relevance. Am J Health Behav. 2003 Nov-Dec;27 Suppl 3:S227-32. doi: 10.5993/ajhb.27.1.s3.6. PMID 14672383
- [Background] Lee DJ, Fleming LE, Arheart KL, LeBlanc WG, Caban AJ, Chung-Bridges K, Christ SL, McCollister KE, Pitman T. Smoking rate trends in U.S. occupational groups: the 1987 to 2004 National Health Interview Survey. J Occup Environ Med. 2007 Jan;49(1):75-81. doi: 10.1097/JOM.0b013e31802ec68c. PMID 17215716
- [Background] Maibach EW, Maxfield A, Ladin K, Slater M. Translating health psychology into effective health communication: the american healthstyles audience segmentation project. J Health Psychol. 1996 Jul;1(3):261-77. doi: 10.1177/135910539600100302. PMID 22011991
- [Background] Nigg CR, Burbank PM, Padula C, Dufresne R, Rossi JS, Velicer WF, Laforge RG, Prochaska JO. Stages of change across ten health risk behaviors for older adults. Gerontologist. 1999 Aug;39(4):473-82. doi: 10.1093/geront/39.4.473. PMID 10495586
- [Background] Okechukwu CA, Krieger N, Sorensen G, Li Y, Barbeau EM. MassBuilt: effectiveness of an apprenticeship site-based smoking cessation intervention for unionized building trades workers. Cancer Causes Control. 2009 Aug;20(6):887-94. doi: 10.1007/s10552-009-9324-0. Epub 2009 Mar 20. PMID 19301135
- [Background] Okechukwu CA, Krieger N, Sorensen G, Li Y, Barbeau EM. Testing hypothesized psychosocial mediators: lessons learned in the MassBUILT study. Health Educ Behav. 2011 Aug;38(4):404-11. doi: 10.1177/1090198110380544. Epub 2011 Apr 7. PMID 21474634
- [Background] Perry RJ, Keller PA, Fraser D, Fiore MC. Fax to quit: a model for delivery of tobacco cessation services to Wisconsin residents. WMJ. 2005 May;104(4):37-40, 44. PMID 16117232
- [Background] Ringen K, Anderson N, McAfee T, Zbikowski SM, Fales D. Smoking cessation in a blue-collar population: results from an evidence-based pilot program. Am J Ind Med. 2002 Nov;42(5):367-77. doi: 10.1002/ajim.10129. PMID 12382249
- [Background] Slater MD. Theory and method in health audience segmentation. J Health Commun. 1996 Jul-Sep;1(3):267-83. doi: 10.1080/108107396128059. PMID 10947364
- [Background] Smith DR. Tobacco smoking by occupation in Australia and the United States: a review of national surveys conducted between 1970 and 2005. Ind Health. 2008 Jan;46(1):77-89. doi: 10.2486/indhealth.46.77. PMID 18270453
- [Background] Sorensen G, Emmons K, Hunt MK, Barbeau E, Goldman R, Peterson K, Kuntz K, Stoddard A, Berkman L. Model for incorporating social context in health behavior interventions: applications for cancer prevention for working-class, multiethnic populations. Prev Med. 2003 Sep;37(3):188-97. doi: 10.1016/s0091-7435(03)00111-7. PMID 12914824
- [Background] Sorensen G, Barbeau E, Hunt MK, Emmons K. Reducing social disparities in tobacco use: a social-contextual model for reducing tobacco use among blue-collar workers. Am J Public Health. 2004 Feb;94(2):230-9. doi: 10.2105/ajph.94.2.230. PMID 14759932
- [Background] Sorensen G, Barbeau EM, Stoddard AM, Hunt MK, Goldman R, Smith A, Brennan AA, Wallace L. Tools for health: the efficacy of a tailored intervention targeted for construction laborers. Cancer Causes Control. 2007 Feb;18(1):51-9. doi: 10.1007/s10552-006-0076-9. PMID 17186421
- [Background] Velicer WF, DiClemente CC, Prochaska JO, Brandenburg N. Decisional balance measure for assessing and predicting smoking status. J Pers Soc Psychol. 1985 May;48(5):1279-89. doi: 10.1037//0022-3514.48.5.1279. PMID 3998990
- [Background] Vladutiu CJ, Nansel TR, Weaver NL, Jacobsen HA, Kreuter MW. Differential strength of association of child injury prevention attitudes and beliefs on practices: a case for audience segmentation. Inj Prev. 2006 Feb;12(1):35-40. doi: 10.1136/ip.2004.007153. PMID 16461418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We invited 1937 union members to participate; 1638 members completed the baseline survey (84.6%). Of those, 553 were current smokers, 1066 were non-smokers, and the smoking status was unknown for 19 individuals. The smoking rate was 33.8%, slightly lower than expected based on previous studies in this population.
Pre-assignment Details: Of 553 current smokers, 111 were not eligible for study inclusion because they either did not sign a consent form (n=49), were not eligible for union benefits (n=57), or had too much data missing at baseline (n=5). The 442 eligible smokers were separated into the four segments and then randomized into the intervention group or the control group.
Groups:
- Intervention Group: Targeted messaging
  Targeted messaging: 1 informational letter plus 6 targeted mailed messages and 6 booster text messages
  Standard messaging: 1 informational letter
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 223 | 219
Completed | 170 | 175
Not Completed | 53 | 44
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 35 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 223 | 219 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.64 (11.54) | 35.18 (11.54) | 35.33 (11.44)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 221 | 218 | 439
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 220 | 218 | 438
Region of Enrollment [Number; unit: participants]
  United States | 223 | 219 | 442

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in Smoking Cessation Program
Description: Enrollment records from the union-sponsored smoking cessation program
Time Frame: up to 12 months after recruitment
Population: Includes all study subjects
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 223 | 219
participants | 5 | 4
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.76, Chi-squared

2. Secondary Outcome: Quit Smoking
Description: At follow-up, subjects will report current smoking status. ("Do you currently smoke (have you smoked in the last 30 days)?" [Yes, I smoked within the past 30 days; No, but I have smoked in the past 6 months; No, and I have not smoked in more than 6 months]). We will report the % of subjects who have not smoked in the last 30 days and will compare the intervention group with the control group.
Time Frame: 7 months after baseline
Population: Secondary outcomes were collected via self-report survey approximately 7 months after study enrollment; 345 subjects (78%) completed the follow-up survey.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 170 | 175
percentage of participants | 17.1 | 16.0
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.79, Regression, Logistic

3. Secondary Outcome: Changes in Smoking Behaviors (Frequency and Quantity)
Description: At baseline and follow-up, subjects will report smoking frequency ("How often do you smoke?" [everyday, at least 4 days/week, 1-3 days/week, less than one day/week]) and quantity ("On days that you smoke, how many cigarettes do you have per day?" [10 or less, 11-20, 21-30, 31 or more]). We will report the % of subjects who smoke less frequently and smoke fewer cigarettes per day at follow-up compared to baseline. We will compare the intervention group with the control group.
Time Frame: 7 months after recruitment
Population: Secondary outcomes were collected via self-report survey approximately 7 months after study enrollment; 345 subjects (78%) completed the follow-up survey. This outcome was only measured in those who reported smoking in the last 30 days (n=288, 83.5%).
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 141 | 147
percentage of participants
  Smoked less frequently | 14.8 | 12.2
  Smoked fewer cigarettes per day | 24.8 | 19.7
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Smoking frequency; Test type: Superiority or Other; p = 0.63, Regression, Logistic
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Smoking quantity; Test type: Superiority or Other; p = 0.30, Regression, Logistic

4. Secondary Outcome: Changes in Readiness to Quit Smoking in the Next 6 Months
Description: Subjects will answer the following question at both baseline and follow-up surveys: "Are you seriously considering quitting smoking in the next 6 months?" [yes/no]. We will report % of subjects who said "no" at baseline and "yes" at follow-up to determine changes in readiness to quit smoking and compare between intervention and control groups.
Time Frame: 7 months after recruitment
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 141 | 147
percentage of participants | 9.2 | 13.6
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.28, Regression, Logistic

5. Secondary Outcome: Changes in Motivation to Quit Smoking and Thinking About Quitting Smoking
Description: At baseline and follow-up, subjects will answer questions about motivation to quit smoking ("How motivated are you to quit smoking at this time? [scale: 1 (not at all) - 10 (extremely)]) and thinking about quitting smoking ("Each rung on this ladder represents where various smokers are in their thinking about quitting. Circle the number that indicates where you are now. [0 (no thoughts of quitting) -10 (taking action to quit)]). We will report the % of subjects who reported more motivation to quit and greater thinking about quitting at follow-up compared to baseline. We will compare the intervention group with the control group.
Time Frame: 7 months after recruitment
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 141 | 147
percentage of participants
  More motivated to quit smoking | 14.9 | 23.8
  Greater thinking about quitting smoking | 12.1 | 22.5
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Motivation to quit; Test type: Superiority or Other; p = 0.09, Regression, Logistic
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Thinking about quitting; Test type: Superiority or Other; p = 0.04, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/219
Other Adverse Events (participants affected / at risk) | 0/223 | 0/219

LIMITATIONS AND CAVEATS:
Messages were based on feedback from a small sample that over-represented young workers; messages may not have been applicable to all union members. Intervention reach was low; only 42% of intervention participants reporting receiving postcards.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No